CLINICAL TRIAL: NCT02789202
Title: Efficacy, Cost-efficacy and Parental Acceptability of Using Diammine Silver Fluoride in Arresting Enamel Caries Lesions on Babies' Occlusal Surfaces
Brief Title: Diammine Silver Fluoride in Arresting Enamel Caries Lesions on Babies' Occlusal Surfaces
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Sao Paulo (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, Mariana Minatel Braga, PhD, Associate professor, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SDFtrials-03
Record Dates: First submitted 2016-05-25; First posted 2016-06-02 (Estimated); Last update posted 2018-03-21 (Actual); Status verified 2018-03

CONDITIONS: Dental Caries
Keywords: dental caries; deciduous tooth
MeSH Terms: conditions — Dental Caries | interventions — silver diamine fluoride; Sodium Fluoride

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Silver Diamine Fluoride (Experimental): Control treatment
  Interventions: Other: Silver diamine fluoride
- Fluoride Varnish (Active Comparator): Test treatment
  Interventions: Other: Fluoride Varnish

INTERVENTIONS:
Other: Silver diamine fluoride — Treatment of initial dental caries lesion in occlusal surface using the silver diamine fluoride.
  Other Names: SDF
  Arms: Silver Diamine Fluoride
Other: Fluoride Varnish — Treatment of initial dental caries lesion in occlusal surface using the fluoride varnish
  Other Names: sodium fluoride
  Arms: Fluoride Varnish

SUMMARY:
This study aims to verify the actual possibility of using silver diammine fluoride (SDF) in arresting enamel caries lesions on occlusal surfaces of primary molars in babies. Besides, the cost-efficacy and also parental acceptability of using SDF will be evaluated. For this, 100 babies 1-3 years will be examined and treated in a mobile dental unit, which will temporarily be parked in public schools of Barueri, Sao Paulo, Brazil. The caries diagnosis will be conducted using the International Caries Detection and Assessment System (ICDAS). Babies with initial lesions will be randomized concerning the treatment in Group A (SDF) and Group B (fluoride varnish). Participants will be examined in the baseline and followed by 6, 12, 18 and 24 months. As primary outcome, caries progression into dentine will be considered. Acceptability reported by parents after treatments, the time and estimated money spent for treating will also be collected. Social and biological data that could be related to efficacy of techniques will be also collected. Multilevel analyses will be performed to check which technique will be most effective and possible factors associated to its efficacy. Discomfort, acceptability and costs will be compared between/among the approaches used to arrest enamel caries lesions.

ELIGIBILITY:
Inclusion Criteria:

* Babies 1 to 3 years;
* Babies with initial dental caries lesion.

Exclusion Criteria:

* Parents who do not consent.

Ages: 1 Year to 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2014-10; Primary Completion 2018-12 (Estimated); Study Completion 2020-08 (Estimated)

PRIMARY OUTCOMES:
Number of caries lesions which progressed to dentine | 24 months
  Assessment of caries lesions severity in order to identify those which progressed to dentine (ICDAS scores 4 to 6)

SECONDARY OUTCOMES:
Parental acceptability to the treatment using a VAS scale | 12 months
  Parents will be asked to report their satisfaction with the treatment using a VAS scale

OTHER OUTCOMES:
Direct and Indirect Costs of initial procedures and consequent interventions during 24 months | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Mariana Minatel Braga, PhD, Principal Investigator — University of Sao Paulo
Locations (1):
- University of São Paulo, São Paulo, Brazil